CLINICAL TRIAL: NCT04098939
Title: Replaceability of Fluoroscopy and Ultrasound in the Evaluation of Hemidiaphragm Excursion"
Brief Title: Replaceability of Fluoroscopy and Ultrasound in the Evaluation of Hemidiaphragm Excursion
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Diaphragm Study AUH
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-03

CONDITIONS: Diaphragm Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants undergoing ultrasound and fluoroscopy assessment of diaphragm excursion.
  Interventions: Diagnostic Test: Diaphragm evaluation

INTERVENTIONS:
Diagnostic Test: Diaphragm evaluation — Ultrasound and radiographic evaluation of diaphragm function

SUMMARY:
Precise measurement of diaphragm function is difficult. Several methods exist. No are sufficiently validated.

With this study, the investigators wish to investigate the validity of different ultrasound and radiological methods and compare them with inspiratory pressure measurements.

DETAILED DESCRIPTION:
Fluoroscopy assessment of diaphragm motility is obtained and simultaneously correlated to sonographic assessments of motility.

ELIGIBILITY:
Inclusion Criteria:

* Completed informed consent
* one of the following conditions:

  * Healthy participants, control group
  * Lung disease group.

    * COPD or
    * Ideopatic pulmonary fibrosis.
  * Heart disease group.

Heart disease that lead to:

* heart transplantat or
* left ventricular assist device.

Exclusion Criteria:

* Known diaphragm dysfunction.
* Neuromuscular disease.
* Pleural effusion.
* Pneumothorax.
* In the healthy group: Significant comorbidity that affect heart og lung function (arterial hypertention, mild valve disease and COPD without symptoms are accepted).
* In the healthy group and in the lung disease group: Previous thorax surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants. Participants with prior COVID-19 infection. Participants with lung diseases. Participants with heart diseases.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren H Skaarup, Study Chair — Aarhus University Hospital; Peter Juhl-Olsen, Study Chair — Aarhus University Hospital; Brian Løgstrup, Study Chair — Aarhus University Hospital; Thomas Birkelund, Study Chair — Aarhus University Hospital; Morten Bendixen, Study Chair — Aarhus University Hospital
Locations (1):
- Søren Helbo Skaarup, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Height, cm [Mean (Standard Deviation); unit: Centimeters] | 176.7 (10.8)
Weight. Kg [Mean (Standard Deviation); unit: kilograms] | 81.9 (17.4)

OUTCOME MEASURES:

1. Primary Outcome: Diaphragm Function
Description: Movement of diaphragm measured with ultrasound Ultrasound measures: Diaphragm excursion in centimeters with M-mode.
Time Frame: during intervention, up to 1 hour
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Participants
Number analyzed (Participants) | 42
centimeters | 4.25 (2.05)
Statistical Analysis 1: Comparison: Participants; Test type: Equivalence — Bland-Altman plots; p < 0.05, Bland-Altman plots — Analysis of Bland-Altman plots; Analysis of Bland-Altman plots; Bland-Altman plots = 0.39, 95% CI 2-sided [0.26 to 1.04]; Analysis of Bland-Altman plots

ADVERSE EVENTS:
Time Frame: Immediate after intervention, up to one hour.
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04098939/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT04098939/ICF_001.pdf